CLINICAL TRIAL: NCT03078777
Title: The Effect Dialysis on the Pharmacokinetics of Fexofenadine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 108170
Record Dates: First submitted 2017-03-07; First posted 2017-03-13 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Hemodialysis
Keywords: Pharmacokinetics
MeSH Terms: interventions — fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Dialysis (Experimental): Patients will take 120 mg of fexofenadine three hours prior to dialysis and plasma concentration measured three hours following dosing.
  Interventions: Drug: Fexofenadine
- Post-Dialysis (Experimental): Patients will take 120 mg of fexofenadine at the end of their dialysis session and plasma concentration measured three hours following dosing.
  Interventions: Drug: Fexofenadine

INTERVENTIONS:
Drug: Fexofenadine — Fexofenadine will be administered to patients.

SUMMARY:
The Investigators recently completed and published a study that demonstrated that fexofenadine pharmacokinetics are significantly altered in dialysis patients (Thomson et al. (2015) American Journal of Kidney Diseases 65(4):574-582). In this study, patients were studied directly before routine dialysis treatment. Other published literature suggests the timing of the dose of some drugs (before or after dialysis) may have a profound impact on the drug pharmacokinetics (Nolin et al (2006) 17(9):2363-7). The hypothesis is that compounds that accumulate in the blood of patients with kidney failure impact the pharmacokinetics such that dosing before or after dialysis produces significantly different blood levels of the drug.

DETAILED DESCRIPTION:
This will be an open, randomized pharmacokinetic study in 30 patients treated by dialysis. Patients will be asked to spend an additional 3 hours at the hospital on each of two study days separated by at least a week. At the first study visit, the patient will be randomized to receive the drug fexofenadine (120 mg, orally) either 3 hour prior to, OR at the conclusion of their regularly scheduled dialysis treatment. Three hours following fexofenadine administration, a single 4 mL (approximately 1 teaspoon) blood sample will be drawn. One week or more after the first study day, the patient will have the study repeated but with the timing of the dose altered to match the randomization. For example, if at the first study visit the patient received fexofenadine after their dialysis session, they will now receive the drug 3 hours prior to their dialysis session. The blood sample will be centrifuged immediately and plasma stored at -80 celsius until analysis. Fexofenadine concentration will be determine by liquid chromatography coupled to mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by any dialysis modality (e.g. hemodialysis, peritoneal dialysis) for at least 90 days prior to study enrolment.

Exclusion Criteria:

* Current or recent (within two weeks) hepatic or gastrointestinal morbidity. Inability or refusal to provide written informed consent. Unable to provide a blood sample. Female patients that are pregnant will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-29 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Plasma Fexofenadine Concentration | 3 hours following dosing
  Measurement of Plasma Fexofenadine Concentration

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No